CLINICAL TRIAL: NCT06255197
Title: Characteristics, Treatment Patterns and Outcomes for Patients With Surgically Resected Lung Cancers
Status: Recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: LungReal_01
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Lung Adenocarcinoma; Lung Squamous Cell Carcinoma; Non Small Cell Lung Cancer; Small-cell Lung Cancer
Keywords: Lung cancer; Surgery; Real world
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with surgically resected lung cancer: Patients who were diagnosed with lung cancer and received surgical resection in participating medical centers during the designed study period.

SUMMARY:
This study is a multi-center, observational, real-world study for patients with resected lung cancers in China. With the help of a properly designed data processing algorithm and extensively performed data quality assurance, this study aims to harness the potential of real-world big data to (1) describe characteristics and treatment patterns and their evolving trends; (2) discover features associated with overall survival; and (3) address recently-emerging clinical questions.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related deaths in China. The recent decade witnessed rapid evolving of demographics, pathological features and prognoses of patients with surgically resected lung cancers. The introduction of minimally invasive surgery (MIS) concept and techniques, targeted therapy and immunotherapy changed treatment landscape for patients with surgically resected lung cancers. With more early-stage lung cancers discovered due to the application of CT screening, questions focusing on extent of lung resection, lymph node dissection, application of targeted or immune-therapy to early-stage lung cancers are emerging. This study aims to create a cohort of patients with surgically resected lung cancers and an analytic framework to address the aforementioned clinical questions.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18.
* Have received surgical resection for lung malignancies.

Exclusion Criteria:

* Participants whose data are of low quality, poor completeness or poor internal linkage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants eligible for this study would be screened from consecutive patients who received surgical resection for lung malignancies in participating medical centers during the designed study period.
Sampling Method: Non-Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | January 2014 to December 2031
  Time from surgery to death from any cause.

SECONDARY OUTCOMES:
Baseline characteristics of included participants | January 2014 to December 2028
  Demographics, symptoms at diagnosis, tobacco exposure, family history, previous medical history, etc.
Treatment patterns of included participants | January 2014 to December 2028
  Extent of lung resection and lymph node dissection, application of certain surgical techniques or not; application of chemotherapy, targeted therapy, immunotherapy and/or radiotherapy before and/or after surgery.
Pathological characteristics of included participants | January 2014 to December 2028
  Location, size, classification, presence or absence of certain pathological features of resected tumor(s); number of metastasized and dissected lymph nodes in each station.
Features associated with overall survival | First analysis is anticipated to be performed from April to August 2024; the final analysis is anticipated in 2032.
  Features within the range of collected baseline characteristics, treatment patterns and pathological characteristics that are associated with overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, MD-PhD, Principal Investigator — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, CAMS and PUMC
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No